CLINICAL TRIAL: NCT03865615
Title: The Effects of Intranasal Oxytocin on Approach Bias and Craving in Moderate to Heavy Alcohol Drinkers
Brief Title: Oxytocin on Approach Bias and Craving
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID made study visits impossible during the funding period.
Sponsor: Jennifer Mitchell (Other)
Responsible Party: Sponsor-Investigator, Jennifer Mitchell, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Oxytocin Approach
Record Dates: First submitted 2018-12-21; First posted 2019-03-07 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Within-subject, randomized, placebo-controlled, counterbalanced, crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin First (Experimental): Subjects will receive oxytocin prior to their first scanning session, and placebo prior to their second scanning session.
  Interventions: Drug: Oxytocin; Drug: Placebo
- Placebo First (Experimental): Subjects will receive placebo prior to their first scanning session, and oxytocin prior to their second scanning session.
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — intranasal oxytocin 40IU/mL
  Other Names: Syntocinon
Drug: Placebo — Placebo

SUMMARY:
This will be a laboratory-based investigation of the behavioral and neural effects of intranasal oxytocin on craving for alcohol and approach bias in moderate to heavy alcohol using subjects. This study uses a within-subject, randomized, placebo-controlled, counterbalanced, crossover design to compare the effects oxytocin and placebo. In this way, all subjects will be scanned twice; once following oxytocin administration and once following placebo administration, and will complete a series of behavioral tasks (both in and out of the scanner) at both visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who are 21-40 years of age
* If female, 10 or more alcoholic drinks must be consumed weekly.
* If male, 14 or more alcoholic drinks must be consumed weekly.
* Meets DSM-V criteria for Alcohol Use Disorder (AUD).
* Score 8 or greater on the Alcohol Use Disorders Identification Test (AUDIT)
* If female, must be non-lactating, not pregnant, and using a reliable contraception method (i.e. abstinence, intrauterine device [IUD], hormonal birth control, or barrier method).
* Native English speaker
* Right handed
* High school graduate or equivalent.
* Able and willing to provide an informed consent.
* Able to understand and follow the instructions of the investigator

Exclusion Criteria:

* Positive urine drug screen (except marijuana).
* Using cocaine, stimulants (other than nicotine and caffeine), amphetamines, hallucinogens, ecstasy, opiates, sedatives, pain pills, sleeping pills, or other psychoactive drugs within 2 weeks of the start of the study (except marijuana).
* Marijuana use more than 3 times/week.
* Current enrollment in an alcohol, or other drug treatment program or current legal problems relating to alcohol, or other drug use.
* Currently trying to quit alcohol use.
* History of major alcohol related complications within the preceding 2 years (liver failure/cirrhosis, pancreatitis, esophageal varices, etc.).
* Has a history of atrophic rhinitis, recurrent nose bleeds, cranial surgical procedures, hypophysectomy, chronic congestion, or sinus problems.
* Has a history of cardiac arrhythmia.
* Clinically significant medical or psychiatric illness requiring treatment as determined by screening blood tests, medical history, and/or physical exam performed or reviewed by the study physician.
* Severely low blood (< 90/50) pressure or uncontrolled high blood pressure (>160/100).
* SGPT/ALT or SGOT/AST values greater than 2x upper limit of normal.
* BAC level > 0.00% at the beginning of screening visit (within margin of error of detection).
* Has a neurological dysfunction or psychiatric disorder (confirm with study physician).
* Has a history of brain trauma (confirm with study physician).
* Has an allergy or intolerance to oxytocin.
* Has received an investigational drug within 30 days of Screening Visit.
* Has any MRI scanning contraindications.
* Has a history of claustrophobia.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Alcohol cue craving score | ~ 90 minutes post study drug administration
  Subjects will be asked to perform a standardized alcohol cue exposure paradigm and be asked to rate their subjective craving following alcohol cue presentation using a standard visual analog scale. Craving scores (ranging from 1-10 on VAS) will be compared across both the active study drug and placebo.
Image approach task | ~ 90 minutes post study drug administration
  Subjects will be asked to perform an image approach task where subjects are presented with a series of images and asked to pull or push a joystick following each presentation. Response direction and speed are recorded and compared across both the active study drug and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mitchell, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No